CLINICAL TRIAL: NCT04691986
Title: Impacts of Nicotinamide Riboside on Functional Capacity and Muscle Physiology in Older Veterans
Acronym: NR-VET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University at Buffalo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: E3396-R; RX003396 (Other Grant/Funding Number: VA RR&D Service)
Record Dates: First submitted 2020-12-10; First posted 2020-12-31 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Sarcopenia; Nicotinamide Adenine Dinucleotide Concentration; Muscle Quality and NAD+ Content
Keywords: muscle; strength; endurance; gait speed; grip strength; frailty; muscle fibers; mitochondria; inflammation; resilience; aging
MeSH Terms: conditions — Sarcopenia; Frailty; Inflammation | interventions — nicotinamide-beta-riboside

STUDY DESIGN:
Intervention Model Description: The study will be conducted as a double-blind randomized controlled trial. Participants will be randomly assorted to receive either the nicotinamide riboside supplementation or a placebo pill.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The study design participants, care providers, and investigators will be blinded to the group designation of the participants. To accomplish this, the study statistician will coordinate with the VA pharmacy to assign groups to participants and to dispense appropriate treatments to the study coordinator to give to study participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NR Supplementation (Experimental): Participants in this group will receive NR supplementation at 1000 mg per day (given as 2x250mg capsules morning and 2x250mg at night).
  Interventions: Dietary Supplement: Nicotinamide Riboside
- Placebo supplementation (Placebo Comparator): Participants in this group will receive placebo given as 2 pills in the morning and 2 pills at night. Placebo pills contain micro cellulose which is likewise found in NR containing capsules.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Nicotinamide Riboside — Nicotinamide Riboside is a form of vitamin B3 and is naturally occurring in humans.
  Other Names: NR
  Arms: NR Supplementation
Other: Placebo — Placebo pills contain micro cellulose powder.
  Arms: Placebo supplementation

SUMMARY:
Frailty is an age-associated clinical condition of poor physiological reserve that increases risks for falls, hospitalization and mortality. Nicotinamide adenine dinucleotide (NAD) is a critical co-factor needed for many cellular processes. The natural levels of NAD decline aging and this has been linked to physical performance decline in animals. Human trials have demonstrated that nicotinamide riboside (NR), a form of vitamin B3, is safe and effectively increases NAD+ levels. In animal studies, NR improves treadmill performance and muscle quality. Here the investigators propose a double-blind randomized control trial to assess the benefits of NR supplementation on human muscle function and physiology. The investigators anticipate the research findings will support the use of this nutritional supplement to improve the health of Veterans during aging.

DETAILED DESCRIPTION:
Frailty is increasingly seen within the aging population and is driven largely by musculoskeletal declines. Nearly 9 million Veterans are now 65 years of age or older with impairments in functional capacity, reduction in quality of life, and an increase in the use of health care services and associated costs. An estimated 45-50% of those over the age of 85 are frail, which could represent well over 1 million Veterans. Aging, which significantly contributes to frailty, is highly correlated with reduced levels of nicotinamide adenine dinucleotide (NAD+), an essential mediator in mitochondrial function. Restoration of cellular NAD+ levels is gaining support as a therapeutic strategy to maintain and even enhance functional capacity during aging. Nicotinamide riboside (NR) - an NAD+ precursor - enhances physical activity and mitochondrial health in mice. Furthermore, NR was recently shown to be safe in human clinical trials for boosting NAD+, yet the benefits for human physical performance and muscle physiology are unknown. Therefore, the goal of this project is to establish a double-blind randomized control trial to assess the impacts of NR on functional capacity, muscle function and structure, and mRNA signaling in healthy older adults. Towards this goal, this study will investigate healthy older individuals between the ages of 65 and 85 who will receive NR or a placebo for a period of 3 months. Participants will be tested for frailty, gait speed, and muscle strength at each time point. Additionally, muscle biopsies and serum will be collected to assess changes in muscle fiber histology, mitochondrial biomass and activity, and mRNA profiles. This project will provide greater insight into NR supplementation as a therapeutic strategy to stave off frailty and maintain resilience during aging.

ELIGIBILITY:
Inclusion Criteria:

* Ages 65-85
* Male or female
* Any race
* Ability to use an exercise bike
* Medically cleared for muscle biopsy

Exclusion Criteria:

* Severe Co-morbidity

  * examples include, but not limited to:
  * congestive heart failure class equal to or above III
  * chronic obstructive pulmonary disorder (COPD) gold stage IV
  * chronic kidney disease equal to or above stage
* A VA-SLUMS cognitive screen score of less than or equal to 20
* Body mass index greater than or equal to 40

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Sub-maximal oxygen uptake test (VO2max) | Change from baseline to endpoint at 12 weeks
  Participants are asked to exercise on an recumbent exercise bike as the resistance increases over time. During the exercise, participants are asked to breath through a mask that is connected to a oxygen and carbon dioxide measuring device. Participant will be asked to continue until they report exhaustion, reach 85% of heart rate maximum, or if there are medical concerns. The assessment last for approximately 15 minutes and provides data the pertain to an individuals lung capacity, breathing rate, and endurance.
Muscle strength | Change from baseline to endpoint at 12 weeks
  Leg and arm strength will be measured using a small handheld dynamometer where the device is placed on the wrist or ankle as the participant is asked to extend or contract the limb with full force.
Gait speed | Change from baseline to endpoint at 12 weeks
  Participants are asked to perform a timed walk of approximately 15 feet in length

SECONDARY OUTCOMES:
Frailty assessment | Change from baseline to endpoint at 12 weeks
  Frailty is a syndrome marked by greater susceptibility to adverse outcomes like falls and disability. Frailty diagnosis in this study is conducted as having 3 or more of the following risk factors - unexpected weight loss in a 1 year time frame, weak grip strength measured by a hand dynamometer device, slow gait speed in a 15 foot walk test, low activity levels assessed with a survey question, and poor endurance also assessed by a survey question.
Short Physical Performance Battery | Change from baseline to endpoint at 12 weeks
  The Short physical performance battery (SPPB) is a battery of test often used in geriatric research to capture functional capacity in older adults. The test includes a balance and coordination assessment via asking participants to hold stances with different foot positions, a gait speed test of approximately 8 feet, and a chair rise timed test where a participant is asked to rise from a chair 5 times.
Quality of life assessment | Change from baseline to endpoint at 12 weeks
  Quality of life assessment is performed using the Quality of life, enjoyment, and satisfaction questionnaire - short form (Q-LES-Q-SF) survey instrument. The survey instrument scores from 0 to 70 with a greater score representing better quality of life.
Cognitive screen | Change from baseline to endpoint at 12 weeks
  Cognitive status will be assessed using the VA - St. Louis University Mental Survey (VA-SLUMS) involving memory tests, shape recognition, and story recall. The survey scores range from 0-30, with a higher score representing greater cognitive capability.
Serum inflammatory biomarkers | Change from baseline to endpoint at 12 weeks
  Chronic inflammation may be indicative of distress and lead to chronic diseases. The study will examine changes in inflammatory markers, C-reactive protein, interleukin-6, and interleukin-10.
Body Composition (Lean and fat mass) | Change from baseline to endpoint at 12 weeks
  Body composition will be measured using bioelectric impedance (BIA) - a technique where participants are asked to stand on the measurement device and hold on to two metal handles. A light - and non-detectable - current is then transmitted allowing for collection of body fat and lean mass in the subject. The assessment takes roughly 2-3 minutes.
Blood occlusion resilience | Change from baseline to endpoint at 12 weeks
  The assessment is a measurement of the decline and restoration of blood oxygenation in the arm in response to the application of a blood pressure cuff to restrict blood flow. Blood oxygenation is measured by a technique called functional near infrared spectroscopy (fNIRS), that requires the placement of a small sensor on the lower forearm. The assessment takes roughly 6-7 minutes.
6-minute walk and heart rate recovery | Change from baseline to endpoint at 12 weeks
  Participants will be asked to walk continuously at a brisk pace for 6 minutes as a measure of endurance. Additionally, they will be asked to wear a pulse-blood oxygenation monitor that will allow continuous measurement of heart rate. Following the assessment, the participant will be asked to be seated for 5 minutes to measure heart rate recovery. The assessment will take roughly 15 minutes.
Balance resistance | Change from baseline to endpoint at 12 weeks
  Participants will be asked to stand on a BioSway device that measures sway speed (mm/s). They will be asked to hold balance for 45 seconds in four conditions, A) comfortable stance, B) comfortable stance with eyes closed, C) Narrow stance, and D) Narrow stance with eyes closed. The assessment will take roughly 5 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth L Seldeen, PhD, Principal Investigator — Kansas City VA Medical Center, Kansas City, MO
Locations (1):
- Kansas City VA Medical Center, Kansas City, MO, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data will be shared in publications and seminars culminating from this study. Additionally, de-identified raw data may be made accessible on a public database for research purposes. Individual participant data will be made available to the participant upon request, with the exception of treatment arm, which can be disclosed at the end of the study to protect blinding of investigators. Individual participant data may also be disclosed to current and future collaborators upon acceptance of a formal request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: individual participant data that is used in publication and/or presentations/seminars may become available during the study or immediately thereafter depending on if the data sufficiently merits dissemination. De-identified raw data associated with a publication, if made accessible, will be made available at the time of publication, otherwise, if not associated with a publication, will be made available at the conclusion of the study (06/30/2026).
Access Criteria: De-identified study data that does not containing protected health information (PHI) will be made accessible upon approval of the study team. Written request should be sent to the principal investigator.